CLINICAL TRIAL: NCT00408993
Title: Duloxetine Versus Placebo in the Treatment of Patients With Diabetic Peripheral Neuropathic Pain in China
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: Boehringer Ingelheim (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10599; F1J-MC-HMEQ(a) (Other: Eli Lilly and Company)
Record Dates: First submitted 2006-12-06; First posted 2006-12-08 (Estimated); Results first posted 2009-06-02 (Estimated); Last update posted 2011-07-26 (Estimated); Status verified 2011-07

CONDITIONS: Diabetic Neuropathies
MeSH Terms: conditions — Diabetic Neuropathies | interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Duloxetine (Experimental): 60 mg every day (QD) (morning or evening), by mouth (PO) for 12 weeks (at week 2, dose can be increased to 120 mg at investigator discretion based on response)
  Interventions: Drug: Duloxetine Hydrochloride
- Placebo (Placebo Comparator): Placebo every day (QD), by mouth (PO) for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine Hydrochloride — 60 mg every day (QD) (morning or evening), by mouth (PO)
  Other Names: LY248686; Cymbalta
  Arms: Duloxetine
Drug: Placebo — Placebo every day (QD), by mouth (PO)
  Arms: Placebo

SUMMARY:
To determine if duloxetine 60mg up to 120mg daily can work in treating pain from Diabetic Neuropathy.

ELIGIBILITY:
Inclusion Criteria:

* Have pain due to bilateral peripheral neuropathy caused by Type I or Type II diabetes with the pain beginning in the feet and present for at least 6 months.
* May not be pregnant and agree to utilize medically acceptable and reliable means of birth control during participation in the study.
* Score of 4 or greater on the Brief Pain Inventory on the 24-hour average pain item.

Exclusion Criteria:

* Glycosylated hemoglobin (A1C) > 12%
* Severe hepatic disease
* History of substance abuse or dependence within the past year, excluding nicotine and caffeine.
* Serious or unstable cardiovascular, hepatic (acute liver injury such as hepatitis or severe cirrhosis), kidney, respiratory, blood disorder, seizure disorder, problems with peripheral vascular disease, or other medical conditions or psychiatric conditions that would hinder your participation or likely to lead to hospitalization during the course of the study.
* Taking monoamine oxidase inhibitor (MAOI) within 14 days of starting the study or the potential need to take during or within 5 days after discontinuation from the study.
* Treatment of fluoxetine within 30 days of starting the study.
* Unstable blood sugar control and uncontrolled or poorly controlled hypertension.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 215 (Actual)
Dates: Start 2006-12; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri from 9AM - 5PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (7):
- China (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Beijing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Changsha
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Harbin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nanjing
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Shanghai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wuhan

REFERENCES:
- [Result] Gao Y, Ning G, Jia WP, Zhou ZG, Xu ZR, Liu ZM, Liu C, Ma JH, Li Q, Cheng LL, Wen CY, Zhang SY, Zhang Q, Desaiah D, Skljarevski V. Duloxetine versus placebo in the treatment of patients with diabetic neuropathic pain in China. Chin Med J (Engl). 2010 Nov;123(22):3184-92. PMID 21163113

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 106 | 109
Completed | 87 | 92
Not Completed | 19 | 17
Not completed — Adverse Event | 15 | 4
Not completed — Protocol Violation | 1 | 6
Not completed — Lack of Efficacy | 1 | 4
Not completed — Withdrawal by Subject | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 106 | 109 | 215
Age Continuous [Mean (Standard Deviation); unit: years] | 58.59 (10.37) | 59.90 (9.52) | 59.25 (9.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 59 | 114
  Male | 51 | 50 | 101
Region of Enrollment [Number; unit: participants]
  China | 106 | 109 | 215
Major Depressive Disorder [Number; unit: participants]
  No | 89 | 88 | 177
  Yes | 17 | 21 | 38
Race/Ethnicity [Number; unit: participants]
  East Asian | 106 | 109 | 215
Type of Diabetes Mellitus [Number; unit: participants]
  Type I Diabetes Mellitus | 3 | 2 | 5
  Type II Diabetes Mellitus | 103 | 107 | 210
Beck Depression Inventory-II Total Score [Mean (Standard Deviation); unit: units on a scale] — A 21-item, patient-completed questionnaire to assess characteristics of depression. Each of the 21 items corresponding to a symptom of depression is summed to give a single score. There is a four-point scale for each item ranging from 0 to 3. Total score of 0-13 is considered minimal range, 14-19 is mild, 20-28 is moderate, and 29-63 is severe.
  units on a scale | 15.97 (10.66) | 15.27 (11.49) | 15.61 (11.07)
Brief Pain Inventory 24-Hour Average Pain Score [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 5.47 (1.31) | 5.52 (1.39) | 5.50 (1.35)
Clinical Global Impressions of Severity Score [Mean (Standard Deviation); unit: units on a scale] — Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients.
  units on a scale | 4.26 (0.76) | 4.38 (0.91) | 4.32 (0.84)
Diabetic Neuropathy History [Mean (Standard Deviation); unit: years]
  Duration of Diabetes | 9.07 (6.32) | 10.21 (6.91) | 9.65 (6.63)
  Duration of Diabetic Neuropathy | 2.13 (2.60) | 2.50 (2.98) | 2.32 (2.80)
  Duration of Diabetic Peripheral Neuropathic Pain | 3.09 (3.11) | 3.34 (3.36) | 3.22 (3.24)
Height [Mean (Standard Deviation); unit: centimeters] | 162.64 (7.72) | 162.12 (7.96) | 162.37 (7.83)
Michigan Neuropathy Screening Instrument [Mean (Standard Deviation); unit: units on a scale] — Assesses degree of neuropathy. Responses to 13 out of 15 items are added to obtain total score. Responses of "yes" to items 1,2,3,5,6,8,9,11,12,14,15 are each counted as one point. A "no" response on items 7 and 13 counts as 1 point. Items 4 and 10 are not included in scoring. Total scores range from 0 (no neuropathy) to 13 (severe neuropathy).
  units on a scale | 4.45 (1.19) | 4.59 (1.19) | 4.52 (1.19)
Weight [Mean (Standard Deviation); unit: kilograms] | 64.06 (10.62) | 63.25 (11.52) | 63.65 (11.07)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Week Endpoint in Brief Pain Inventory 24-hour Average Pain Score
Description: A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
Time Frame: Baseline and 12 weeks
Population: Intention to Treat analysis. Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 104 | 109
units on a scale | -2.69 (0.19) | -2.31 (0.18)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; With 104 patients per arm, the study has at least 85% power to detect a treatment group difference of -1.20 points in baseline to endpoint mean change on the BPI 24-hour average pain score between Duloxetine and Placebo. Sample size determined using a two-sided t-test with alpha=0.05, and assuming a common standard deviation of 2.5 and a discontinuation rate of 25%; Test type: Superiority or Other; p = 0.617, ANCOVA — Treatment effects were evaluated based on a two-sided significance level of 0.05 and interaction effects at 0.10. No adjustments for multiple comparisons were made; Model=Treatment, Pooled Investigator and Baseline

2. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Brief Pain Inventory (BPI) Worst Pain, Least Pain, and Current Pain Severity and Average Interference Scores
Description: Measures severity of pain and interference of pain on function. Each severity of pain (worst, least, and current) scores range from 0 (no pain) to 10 (pain as severe as you can imagine). The 7 separate Interference item scores range from 0 (does not interfere) to 10 (completely interferes) and were averaged to provide a single score (0 to 10).
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 104 | 109
units on a scale
  Worst Pain Score | -3.48 (0.27) | -2.93 (0.26)
  Least Pain Score | -1.69 (0.20) | -1.37 (0.20)
  Pain Right Now Score | -2.72 (0.26) | -1.99 (0.25)
  Average Interference Score | -2.28 (0.21) | -1.88 (0.20)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.070, ANCOVA — P-value for Worst Pain Score; Model=Treatment, Pooled Investigator, Baseline and Major Depressive Disorder status at baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.151, ANCOVA — P-value for Least Pain Score; Model=Treatment, Pooled Investigator, Baseline and Major Depressive Disorder status at baseline
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value for Pain Right Now Score; Model=Treatment, Pooled Investigator, Baseline and Major Depressive Disorder status at baseline
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.077, ANCOVA — P-value for Average Interference Score; Model=Treatment, Pooled Investigator, Baseline and Major Depressive Disorder status at baseline

3. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Clinical Global Impression of Severity
Description: Measures severity of illness at the time of assessment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 103 | 109
units on a scale | -1.24 (0.11) | -0.99 (0.11)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.036, ANCOVA; Model=Treatment, Pooled Investigator, Baseline and Major Depressive Disorder status at baseline

4. Secondary Outcome: Time Course of Change in Patient Global Impression - Improvement Scale
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse).
Time Frame: baseline, over 12 weeks
Population: Intention to Treat analysis. Number of randomized patients with at least one non-missing post-baseline data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 98 | 107
units on a scale
  Week 1 (N=5, N=2) | 3.45 (0.56) | 3.51 (0.88)
  Week 2 (N=98, N=107) | 2.91 (0.09) | 3.23 (0.09)
  Week 4 (N=94, N=101) | 2.57 (0.10) | 2.83 (0.10)
  Week 8 (N=91, N=95) | 2.29 (0.11) | 2.76 (0.11)
  Week 12 (N=87, N=92) | 2.27 (0.11) | 2.58 (0.11)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.955, Mixed Models Analysis — P-value for Visit 3; Repeated Measures: Model=Treatment, Pooled Investigator, Visit, Baseline, baseline MDD status, Treatment*Visit and Baseline*Visit
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.004, Mixed Models Analysis — P-value for Visit 4; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.037, Mixed Models Analysis — P-value for Visit 5; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p < 0.001, Mixed Models Analysis — P-value for Visit 6; [statistical method as in outcome 4, analysis 1]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.028, Mixed Models Analysis — P-value for Visit 7; [statistical method as in outcome 4, analysis 1]

5. Secondary Outcome: Change From Baseline to 12 Week Endpoint in EuroQoL Questionnaire - 5 Dimensions (EQ-5D) (US Based Index Score)
Description: The EQ-5D is an assessment of one's overall health. Consists of 5 items. Patients choose 1 of 3 options that best describe the status of each item. The EQ-5D US based index scores range from -0.11 to 1.0 where a score of 1.0 indicates perfect health. A positive change from baseline indicates health improvement.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 101 | 101
units on a scale | 0.12 (0.02) | 0.10 (0.02)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.207, ANCOVA; Model=Treatment, Pooled Investigator, Baseline and Major Depressive Disorder status at baseline

6. Secondary Outcome: Number of Participants Discontinuing Due to Adverse Events
Time Frame: over 12 weeks
Population: Intention to Treat Analysis. All randomized patients.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 106 | 109
participants | 15 | 4
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.008, Fisher Exact

7. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events Reported in >5% of Either Treatment Group by Time of Dosing (Morning or Evening)
Description: Tolerability of morning versus evening dosing, as assessed by the number of participants with spontaneously reported adverse events.
Time Frame: over 12 weeks
Population: Number of randomized patients in each treatment arm for each dosing group
Measure: Number; unit: participants
Groups:
- Duloxetine - Morning Dosing; Duloxetine - Evening Dosing: 60 mg QD (morning or evening), PO for 12 weeks (at week 2, dose can be increased to 120 mg at investigator discretion based on response)
- Placebo - Morning Dosing; Placebo - Evening Dosing: Placebo QD, PO for 12 weeks
Arm/Group | Duloxetine - Morning Dosing | Duloxetine - Evening Dosing | Placebo - Morning Dosing | Placebo - Evening Dosing
Number analyzed (Participants) | 53 | 53 | 56 | 53
participants
  Abdominal discomfort | 3 | 1 | 2 | 4
  Abdominal distension | 7 | 2 | 4 | 3
  Abdominal pain upper | 0 | 4 | 2 | 0
  Anorexia | 4 | 7 | 1 | 1
  Arthralgia | 1 | 0 | 3 | 2
  Asthenia | 2 | 4 | 0 | 1
  Chest discomfort | 2 | 3 | 1 | 0
  Constipation | 4 | 7 | 5 | 4
  Cough | 2 | 0 | 4 | 1
  Decreased appetite | 0 | 3 | 0 | 1
  Diarrhoea | 4 | 6 | 5 | 1
  Dizziness | 5 | 11 | 9 | 3
  Dry mouth | 2 | 4 | 1 | 2
  Dyslipidaemia | 1 | 3 | 1 | 1
  Dysuria | 5 | 4 | 0 | 1
  Fatigue | 3 | 5 | 2 | 6
  Headache | 4 | 2 | 4 | 2
  Hyperhidrosis | 4 | 5 | 1 | 2
  Hypersomnia | 0 | 2 | 2 | 3
  Hypoglycaemia | 5 | 5 | 3 | 2
  Insomnia | 3 | 2 | 3 | 2
  Lethargy | 6 | 5 | 2 | 2
  Nausea | 14 | 18 | 8 | 5
  Pain | 1 | 1 | 3 | 0
  Palpitations | 7 | 3 | 2 | 3
  Pruritus | 2 | 1 | 4 | 4
  Somnolence | 9 | 8 | 2 | 4
  Stomach discomfort | 4 | 3 | 5 | 0
  Therapeutic response unexpected | 6 | 3 | 6 | 6
  Thirst | 4 | 1 | 0 | 1
  Vomiting | 3 | 3 | 2 | 3

8. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Athens Insomnia Scale 8-item and 5-item
Description: Estimates sleep difficulty. Consists of 8 items rated on a 4-point scale of 0 (no problem at all) to 3 (very serious problem). Total score of the 8-item version (sum of items 1-8) ranges from 0-24, while total score of the 5-item (sum of items 1-5) ranges from 0-15.
Time Frame: Baseline and 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 103 | 109
units on a scale
  5-Item Score | -2.27 (0.31) | -1.97 (0.29)
  8-Item Score | -3.58 (0.47) | -3.31 (0.45)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.364, ANCOVA — P-value for 5-Item Score; Model=Treatment, Pooled Investigator, Baseline and Major Depressive Disorder status at baseline
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.590, ANCOVA — P-value for 8-Item Score; Model=Treatment, Pooled Investigator, Baseline and Major Depressive Disorder status at baseline

9. Secondary Outcome: Vital Signs - Weight
Description: Change from baseline to endpoint in body weight.
Time Frame: Baseline and 12 weeks
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: kilograms
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 104 | 109
kilograms | -0.17 (0.21) | -0.03 (0.21)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.620, ANOVA; Model=Treatment and Pooled Investigator

10. Secondary Outcome: Vital Signs - Pulse Rate
Description: Change from baseline to endpoint in pulse rate.
Time Frame: Baseline and 12 weeks
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 104 | 109
beats per minute | 1.71 (1.06) | 0.32 (1.03)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.324, ANOVA; Model=Treatment and Pooled Investigator

11. Secondary Outcome: Vital Signs - Blood Pressure
Description: Change from baseline to endpoint in systolic and diastolic blood pressure.
Time Frame: Baseline and 12 weeks
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 104 | 109
mm Hg
  Systolic Blood Pressure | -0.48 (1.61) | -1.47 (1.56)
  Diastolic Blood Pressure | 0.45 (0.95) | -0.21 (0.92)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.642, ANOVA — P-value for Systolic Blood Pressure; Model=Treatment and Pooled Investigator
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.601, ANOVA — P-value for Diastolic Blood Pressure; Model=Treatment and Pooled Investigator

12. Secondary Outcome: Statistically Significant Change From Baseline to 12 Week Endpoint in Laboratory Measures - Chloride, High Density Lipoprotein, Sodium, and Triglycerides
Description: Significantly different laboratory values between the two groups in baseline to endpoint changes in chloride, high density lipoprotein, sodium, and triglycerides.
Time Frame: Baseline and 12 weeks
Population: Number of randomized patients with a baseline and at least one non-missing post-baseline value, based on first values at scheduled visits.
Measure: Mean (Standard Deviation); unit: millimole/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 99 | 104
millimole/Liter
  Chloride Baseline | 102.94 (3.07) | 102.87 (2.99)
  Chloride Change to Endpoint | -1.15 (3.60) | -0.20 (2.81)
  High Density Lipoprotein Cholesterol Baseline | 1.30 (0.37) | 1.33 (0.33)
  High Density Lipoprotein Change to Endpoint | 0.03 (0.22) | -0.04 (0.19)
  Sodium Baseline | 143.03 (2.83) | 142.76 (3.00)
  Sodium Change to Endpoint | -1.25 (3.64) | -0.19 (2.72)
  Triglycerides Baseline | 1.76 (1.48) | 1.40 (0.76)
  Triglycerides Change to Endpoint | -0.05 (1.07) | 0.26 (1.00)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.014, ANOVA — P-value for Chloride; Sums of squares from ANOVA on the ranks: Model=Treatment and Pooled Investigator for treatment effects p-value
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.005, ANOVA — P-value for High Density Lipoprotein Cholesterol; Sums of squares from ANOVA on the ranks: Model=Treatment and Pooled Investigator for treatment effects p-value
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.011, ANOVA — P-value for Sodium; Sums of squares from ANOVA on the ranks: Model=Treatment and Pooled Investigator for treatment effects p-value
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.044, ANOVA — P-value for triglycerides; Sums of squares from ANOVA on the ranks: Model=Treatment and Pooled Investigator for treatment effects p-value

13. Secondary Outcome: Statistically Significant Change From Baseline to 12 Week Endpoint in Laboratory Measures - Uric Acid
Description: Significantly different laboratory values between the two groups in baseline to endpoint changes
Time Frame: Baseline and 12 weeks
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: micromole/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 99 | 104
micromole/Liter
  Uric Acid Baseline | 293.24 (72.51) | 283.98 (75.88)
  Uric Acid Change to Endpoint | -7.46 (62.19) | 2.49 (53.29)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Test type: Superiority or Other; p = 0.017, ANOVA; Sums of squares from ANOVA on the ranks: Model=Treatment and Pooled Investigator for treatment effects p-values

ADVERSE EVENTS:
Groups:
- Placebo: Placebo
- Duloxetine 60/120 mg QD: Duloxetine 60/120 mg QD
Arm/Group | Placebo | Duloxetine 60/120 mg QD
Serious Adverse Events (participants affected / at risk) | 2 | 2
Other Adverse Events (participants affected / at risk) | 77 | 85
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Duloxetine 60/120 mg QD
Acute myocardial infarction (Cardiac disorders) | 0/109 (0) | 1/106 (1)
Cardiac failure acute (Cardiac disorders) | 1/109 (1) | 0/106 (0)
Nausea (Gastrointestinal disorders) | 1/109 (1) | 1/106 (1)
Vomiting (Gastrointestinal disorders) | 1/109 (1) | 1/106 (1)
Death (General disorders) | 0/109 (0) | 1/106 (1)
Nasopharyngitis (Infections and infestations) | 1/109 (1) | 0/106 (0)
Cerebral infarction (Nervous system disorders) | 0/109 (0) | 1/106 (1)
Renal impairment (Renal and urinary disorders) | 0/109 (0) | 1/106 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0/109 (0) | 1/106 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected / at risk (number of events):
Term (organ system) | Placebo | Duloxetine 60/120 mg QD
Palpitations (Cardiac disorders) | 5/109 (6) | 10/106 (11)
Abdominal discomfort (Gastrointestinal disorders) | 6/109 (6) | 4/106 (4)
Abdominal distension (Gastrointestinal disorders) | 7/109 (7) | 9/106 (9)
Constipation (Gastrointestinal disorders) | 9/109 (10) | 12/106 (14)
Diarrhoea (Gastrointestinal disorders) | 6/109 (6) | 11/106 (11)
Dry mouth (Gastrointestinal disorders) | 3/109 (3) | 6/106 (7)
Nausea (Gastrointestinal disorders) | 12/109 (15) | 31/106 (33)
Stomach discomfort (Gastrointestinal disorders) | 5/109 (6) | 7/106 (7)
Asthenia (General disorders) | 1/109 (1) | 6/106 (6)
Fatigue (General disorders) | 8/109 (8) | 8/106 (8)
Therapeutic response unexpected (General disorders) | 12/109 (18) | 9/106 (15)
Anorexia (Metabolism and nutrition disorders) | 2/109 (2) | 11/106 (11)
Hypoglycaemia (Metabolism and nutrition disorders) | 6/109 (7) | 10/106 (10)
Dizziness (Nervous system disorders) | 12/109 (12) | 16/106 (19)
Headache (Nervous system disorders) | 6/109 (8) | 6/106 (6)
Lethargy (Nervous system disorders) | 4/109 (4) | 11/106 (12)
Somnolence (Nervous system disorders) | 6/109 (6) | 17/106 (18)
Dysuria (Renal and urinary disorders) | 1/109 (1) | 9/106 (9)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3/109 (3) | 9/106 (11)
Pruritus (Skin and subcutaneous tissue disorders) | 8/109 (8) | 3/106 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days